CLINICAL TRIAL: NCT04217005
Title: Enhancing Functional and Cognitive Performances in People With Amputation and Peripheral Neuropathy Through the Restoration of Sensory Feedback in Real World and Virtual Reality Environments
Brief Title: Enhancing Abilities in Amputees and Patients With Peripheral Neuropathy Through Restoration of Sensory Feedback
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ETH Zurich (Other)
Responsible Party: Principal Investigator, Greta Preatoni, Doctoral fellowship, ETH Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-N-97
Record Dates: First submitted 2019-12-10; First posted 2020-01-03 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Lower Limb Amputation Knee; Lower Limb Amputation Above Knee (Injury); Lower Limb Amputation Below Knee (Injury); Diabetic Peripheral Neuropathy
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): amputees or diabetics receiving intervention
  Interventions: Device: Sensory Feedback

INTERVENTIONS:
Device: Sensory Feedback — Subjects will receive a sensory feedback provided by electrical stimulation

SUMMARY:
Many amputees suffer from Phantom Limb Pain (PLP), a condition where painful perceptions arise from the missing limb. Leg amputees wear prostheses that do not provide any sensory feedback, apart from the stump-socket interaction. Increased physical effort associated with prosthesis use as well as discomfort often lead to rejection of artificial limbs. Additionally, the perception of the missing limb and its brain representation, do not match-up with what amputees see (the prosthesis) and this is made worse by the absence of sensory feedback. Therefore, re-establishing the sensory flow of information between the subject's brain and the prosthetic device is extremely important to avoid this mismatch, which creates inadequate embodiment. This study focuses on improving functional abilities and decreasing PLP in amputees thanks to the use of a system able to generate a sensory feedback (SF), which will be provided with a non-invasive electrical stimulation (ES). First, the possibility of enhancing the performance in different functional tasks thanks to the use of SF will be explored. Furthermore, it will be evaluated if SF enhances the prosthesis embodiment and helps restoring a multisensory integration (visuo-tactile), potentially providing also a pain relief. Once tested this system on amputees, also people with peripheral neuropathy and sensory loss will be recruited. Diabetic patients can suffer from symmetrical polyneuropathy (DSPN), which is a common complication caused by prolonged glucose unbalanced levels that lead to nerve damage. Non-invasive ES has been proposed and used as a therapy to treat the chronic pain conditions. In particular, TENS (transcutaneous electrical nerve stimulation) is a type of non-invasive ES, which is able to activate large diameter afferent fibers. The gate control theory of pain states that these large diameter fibers inhibit central nociceptive transmission with a resultant decrease in pain perception. Therefore, also these patients will be recruited to see whether adding a non-invasive SF can enhance their functional motor abilities while diminishing their pain.

The subjects will perform a pool of the following tasks, depending on their residual abilities: motor tasks (walking on ground level and on stairs), cognitive tasks (dual tasks), subjective evaluation of prosthesis weight and description of sensations from ES.

Some tasks will be performed in Virtual Reality environments with and without an active stimulation.

ELIGIBILITY:
Inclusion Criteria:

* transfemoral amputation or transtibial amputation or knee disarticulation or diabetic peripheral neuropathy
* the subject should be healthy other than the amputation and the diabetic neuropathy and in the range of 18-70 years old
* the subject should be able to comfortably walk, sit and stand alone

Exclusion Criteria:

* cognitive impairment
* pregnancy
* Prior or current psychological diseases such as borderline, schizophrenia, Depression or Maniac Depression
* acquired brain injury with residual impairment
* excessive sensitivity or pain to electrical stimulation with surface electrodes
* cybersickness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-12-13 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Visual Analogue scale for pain throughout the study | one month before the study, 2 weeks before the study, immediately before the intervention, immediately after the intervento, after tasks with and without sensory feedback, 2 weeks after last intervention, 1 month after last intervention
  Subjects will complete VAS scale to measure pain level (from 0 to 10, 10 is worst pain immaginable)
Change between tasks with sensory feedback and with no sensory feedback in Ground Reaction Forces | during motor tasks up to 3 weeks
  GRF will be assessed during motor perfomances of the subjects
Change between tasks with sensory feedback and with no sensory feedback in Centre of Mass and Pressure | during motor tasks up to 3 weeks
  CoM and CoP will be assessed during motor perfomances of the subjects
Change from baseline and between tasks with sensory feedback and with no sensory feedback in Vo2 consumption | during motor tasks up to 3 weeks
  metabolic consumption is going to be measured with mobile spiroergometry and compared after walking with and without sensory feedback
Change from baseline between tasks with sensory feedback and with no sensory feedback in Embodiment | immediately after sessions up to 3 weeks
  Embodiment will be measured with questionnaires (from -3 to +3, +3 totally agrees; two questions are from 1 to 10 (to measure vividness, where 10 is max vividness) and from 1 to 100 (to measure prevalence, where 100 is max duration of the embodiment feeling))
Change between tasks with sensory feedback and with no sensory feedback in Visual Analogue scale for confidence | immediately after sessions up to three weeks
  Subjects will complete VAS scale to measure confidence level (from 0 to 10, where 10 is max confidence)
Change between tasks with sensory feedback and with no sensory feedback in Joint torque | during motor tasks up to three weeks
  kinematic measurement
Change in Proprioceptive drift between different conditions | Immediately after sessions in Virtual Reality up to three weeks
  To measure embodiment subjects will be asked after VR sessions to indicate where they feel their leg without looking at the limb in real world. This is a measure of embodiment.
Change in Telescoping measures between different conditions | Immediately after sessions in Virtual Reality up to three weeks
  To measure embodiment subjects will be asked after VR sessions to indicate how long they feel their leg without looking at the limb in real world. This is a measure of embodiment.

SECONDARY OUTCOMES:
Trinity Amputation and Prosthesis Experiences Scales | Immediately before intervention
  Subjects will fill the TAPES to measure their satisfaction with the prosthesis (Scores range from 5 to 25, with higher scores indicating greater levels of adjustment)
Change in Quality of Life in Neurological Disorders | one week before first session and one week after last session
  QoL will be assessed through questionnaires to see if the intevention had impact on this aspect (All Neuro-QOL banks and scales are scored such that a high score reflects more of what is being measured)
Amputee Mobility Predictor | Immediately before the intervention
  Subjects will perform AMPRO to assess K level (scores range from 0 to 47, correspoding to levels of mobility from 1(K1) to 4(K4), where 4 is the best level of mobility)

CONTACTS AND LOCATIONS:
Locations (1):
- ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbott CA, Malik RA, van Ross ER, Kulkarni J, Boulton AJ. Prevalence and characteristics of painful diabetic neuropathy in a large community-based diabetic population in the U.K. Diabetes Care. 2011 Oct;34(10):2220-4. doi: 10.2337/dc11-1108. Epub 2011 Aug 18. PMID 21852677
- [Background] Archer AG, Watkins PJ, Thomas PK, Sharma AK, Payan J. The natural history of acute painful neuropathy in diabetes mellitus. J Neurol Neurosurg Psychiatry. 1983 Jun;46(6):491-9. doi: 10.1136/jnnp.46.6.491. PMID 6875582
- [Background] Burke MJ, Roman V, Wright V. Bone and joint changes in lower limb amputees. Ann Rheum Dis. 1978 Jun;37(3):252-4. doi: 10.1136/ard.37.3.252. PMID 150823
- [Background] Antfolk C, D'Alonzo M, Rosen B, Lundborg G, Sebelius F, Cipriani C. Sensory feedback in upper limb prosthetics. Expert Rev Med Devices. 2013 Jan;10(1):45-54. doi: 10.1586/erd.12.68. PMID 23278223
- [Background] Oddo CM, Raspopovic S, Artoni F, Mazzoni A, Spigler G, Petrini F, Giambattistelli F, Vecchio F, Miraglia F, Zollo L, Di Pino G, Camboni D, Carrozza MC, Guglielmelli E, Rossini PM, Faraguna U, Micera S. Intraneural stimulation elicits discrimination of textural features by artificial fingertip in intact and amputee humans. Elife. 2016 Mar 8;5:e09148. doi: 10.7554/eLife.09148. PMID 26952132
- [Background] Charkhkar H, Shell CE, Marasco PD, Pinault GJ, Tyler DJ, Triolo RJ. High-density peripheral nerve cuffs restore natural sensation to individuals with lower-limb amputations. J Neural Eng. 2018 Oct;15(5):056002. doi: 10.1088/1741-2552/aac964. Epub 2018 Jun 1. PMID 29855427
- [Background] Chow DH, Cheng CT. Quantitative analysis of the effects of audio biofeedback on weight-bearing characteristics of persons with transtibial amputation during early prosthetic ambulation. J Rehabil Res Dev. 2000 May-Jun;37(3):255-60. PMID 10917257
- [Background] Tan DW, Schiefer MA, Keith MW, Anderson JR, Tyler J, Tyler DJ. A neural interface provides long-term stable natural touch perception. Sci Transl Med. 2014 Oct 8;6(257):257ra138. doi: 10.1126/scitranslmed.3008669. PMID 25298320
- [Background] Dailey DL, Rakel BA, Vance CGT, Liebano RE, Amrit AS, Bush HM, Lee KS, Lee JE, Sluka KA. Transcutaneous electrical nerve stimulation reduces pain, fatigue and hyperalgesia while restoring central inhibition in primary fibromyalgia. Pain. 2013 Nov;154(11):2554-2562. doi: 10.1016/j.pain.2013.07.043. Epub 2013 Jul 27. PMID 23900134
- [Background] Dosen S, Markovic M, Strbac M, Belic M, Kojic V, Bijelic G, Keller T, Farina D. Multichannel Electrotactile Feedback With Spatial and Mixed Coding for Closed-Loop Control of Grasping Force in Hand Prostheses. IEEE Trans Neural Syst Rehabil Eng. 2017 Mar;25(3):183-195. doi: 10.1109/TNSRE.2016.2550864. Epub 2016 Apr 7. PMID 27071179
- [Background] Clippinger FW, Seaber AV, McElhaney JH, Harrelson JM, Maxwell GM. Afferent sensory feedback for lower extremity prosthesis. Clin Orthop Relat Res. 1982 Sep;(169):202-6. PMID 7105581
- [Background] Rognini G, Petrini FM, Raspopovic S, Valle G, Granata G, Strauss I, Solca M, Bello-Ruiz J, Herbelin B, Mange R, D'Anna E, Di Iorio R, Di Pino G, Andreu D, Guiraud D, Stieglitz T, Rossini PM, Serino A, Micera S, Blanke O. Multisensory bionic limb to achieve prosthesis embodiment and reduce distorted phantom limb perceptions. J Neurol Neurosurg Psychiatry. 2019 Jul;90(7):833-836. doi: 10.1136/jnnp-2018-318570. Epub 2018 Aug 12. No abstract available. PMID 30100550
- [Background] Sadeghi H, Allard P, Prince F, Labelle H. Symmetry and limb dominance in able-bodied gait: a review. Gait Posture. 2000 Sep;12(1):34-45. doi: 10.1016/s0966-6362(00)00070-9. PMID 10996295
- [Background] Naschitz JE, Lenger R. Why traumatic leg amputees are at increased risk for cardiovascular diseases. QJM. 2008 Apr;101(4):251-9. doi: 10.1093/qjmed/hcm131. Epub 2008 Feb 16. PMID 18281705
- [Background] Kumar D, Marshall HJ. Diabetic peripheral neuropathy: amelioration of pain with transcutaneous electrostimulation. Diabetes Care. 1997 Nov;20(11):1702-5. doi: 10.2337/diacare.20.11.1702. PMID 9353612
- [Background] Kumar D, Alvaro MS, Julka IS, Marshall HJ. Diabetic peripheral neuropathy. Effectiveness of electrotherapy and amitriptyline for symptomatic relief. Diabetes Care. 1998 Aug;21(8):1322-5. doi: 10.2337/diacare.21.8.1322. PMID 9702441
- [Background] Lotze M, Moseley GL. Role of distorted body image in pain. Curr Rheumatol Rep. 2007 Dec;9(6):488-96. doi: 10.1007/s11926-007-0079-x. PMID 18177603
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Petrini FM, Bumbasirevic M, Valle G, Ilic V, Mijovic P, Cvancara P, Barberi F, Katic N, Bortolotti D, Andreu D, Lechler K, Lesic A, Mazic S, Mijovic B, Guiraud D, Stieglitz T, Alexandersson A, Micera S, Raspopovic S. Sensory feedback restoration in leg amputees improves walking speed, metabolic cost and phantom pain. Nat Med. 2019 Sep;25(9):1356-1363. doi: 10.1038/s41591-019-0567-3. Epub 2019 Sep 9. PMID 31501600
- [Background] Petrini FM, Valle G, Bumbasirevic M, Barberi F, Bortolotti D, Cvancara P, Hiairrassary A, Mijovic P, Sverrisson AO, Pedrocchi A, Divoux JL, Popovic I, Lechler K, Mijovic B, Guiraud D, Stieglitz T, Alexandersson A, Micera S, Lesic A, Raspopovic S. Enhancing functional abilities and cognitive integration of the lower limb prosthesis. Sci Transl Med. 2019 Oct 2;11(512):eaav8939. doi: 10.1126/scitranslmed.aav8939. PMID 31578244
- [Background] Crea S, Edin BB, Knaepen K, Meeusen R, Vitiello N. Time-Discrete Vibrotactile Feedback Contributes to Improved Gait Symmetry in Patients With Lower Limb Amputations: Case Series. Phys Ther. 2017 Feb 1;97(2):198-207. doi: 10.2522/ptj.20150441. No abstract available. PMID 28204796
- [Background] Bruce D, Hunter M, Peters K, Davis T, Davis W. Fear of falling is common in patients with type 2 diabetes and is associated with increased risk of falls. Age Ageing. 2015 Jul;44(4):687-90. doi: 10.1093/ageing/afv024. Epub 2015 Mar 3. PMID 25739747
- [Derived] Borda L, Gozzi N, Preatoni G, Valle G, Raspopovic S. Automated calibration of somatosensory stimulation using reinforcement learning. J Neuroeng Rehabil. 2023 Sep 26;20(1):131. doi: 10.1186/s12984-023-01246-0. PMID 37752607